CLINICAL TRIAL: NCT03710486
Title: Vedolizumab and Anti-TNFs Outcomes in Real-World Biologic Ulcerative Colitis and Crohn's Disease Patients
Brief Title: A Study to Observe Vedolizumab and Anti-tumour Necrosis Factors (Anti-TNFs) Outcomes in Real-world Biologic Ulcerative Colitis (UC) and Crohn's Disease (CD) Participants
Acronym: EVOLVE-IBERIA
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Vedolizumab-5047; U1111-1218-0768 (Registry Identifier: WHO); TAK-VDZ-2018-01 (Other: Spanish Agency for Medicine and Health Products)
Record Dates: First submitted 2018-10-16; First posted 2018-10-18 (Actual); Results first posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2023-12

CONDITIONS: Colitis, Ulcerative; Crohn Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Vedolizumab: Participants diagnosed with UC or CD, who have initiated vedolizumab treatment between January 2017 until date of site initiation from the 25 participating sites will be observed from the date of UC or CD diagnosis until one day prior to the date of index vedolizumab treatment initiation during the eligibility period, and then from date of index vedolizumab treatment initiation until the earliest of 6 months (post-index treatment discontinuation, death of participant, lost-to-follow up, or date of chart abstraction). Index date is defined as the date when vedolizumab treatment was initiated.
- Cohort 2: Other Biologic: Participants diagnosed with UC or CD, who have initiated other biologic treatment (infliximab, adalimumab, or golimumab [UC only]) between January 2017 until date of site initiation from the 25 participating sites will be observed from the date of UC or CD diagnosis until one day prior to the date of index other biologic treatment initiation during the eligibility period, and then from date of index other biologic treatment initiation until the earliest of 6 months (post-index treatment discontinuation, death of participant, lost-to-follow up, or date of chart abstraction). Index date is defined as the date when other biologic treatment was initiated.

SUMMARY:
The purpose of this study is to describe treatment patterns associated with first-line and second line biologic use (vedolizumab or other biologic) and to describe the real-world clinical effectiveness of the use (first-line and second line) vedolizumab versus other biologics at least 6 months post-treatment initiation.

DETAILED DESCRIPTION:
This is a retrospective, non-interventional study of participants with CD or UC. The study will review the medical charts of participants who have initiated the first or second line treatment with vedolizumab or another biologic agent (infliximab, adalimumab, or golimumab [UC only]) (index event) during the eligibility period to evaluate the treatment effectiveness, treatment patterns, health care utilization and safety of vedolizumab, and to provide the real-world treatment landscape with anti-TNF alpha therapies.

The study will enroll approximately 400 participants, with 200 participants in each treatment cohort. All participants will be enrolled into two observational groups:

* Cohort 1: Vedolizumab
* Cohort 2: Other Biologics

The data for participants will be collected in two main periods:

* Pre-index Event Period: From the data of diagnosis of UC/CD until one day prior to the date when vedolizumab or other biologic treatment was initiated during the eligibility period.
* Post-index Event Period: From the date when vedolizumab or other biologic treatment was initiated during the eligibility period until the earliest of 6 months (post-index treatment discontinuation, death of participants, lost-to-follow up, or date of chart abstraction initiation.

This multi-center trial will be conducted in Spain and Portugal. The overall time for data collection in the study will be approximately 12 months and the overall duration of the study is approximately 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Has a diagnosis of moderate to severe UC or CD documented in the medical chart.
2. Received at least one dose of vedolizumab or other biologic (infliximab, adalimumab, or golimumab [UC only]) during the eligibility period.
3. Received the biologic treatment as first-line or second line biologic for UC or CD.
4. Has a minimum of six months of follow-up between date of starting biologic therapy (index event) and the date of completion of the participant pre-selection registry.

Exclusion Criteria:

1. Received vedolizumab or another biologic as part of an interventional clinical trial ever in their lifetime (includes index treatment).
2. Index treatment was another biologic therapy other than vedolizumab, infliximab, adalimumab, or golimumab (UC only).
3. Initiated index treatment as combination therapy with two biologic agents.
4. The biologic was prescribed for treatment of perianal disease.
5. Received biologic therapy before the index period for a disease other than inflammatory bowel disease.
6. Medical chart is unavailable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with moderate to severe UC or CD, and have initiated first or second line treatment with vedolizumab and other biologics between January 2017 and the date of site initiation.
Sampling Method: Non-Probability Sample
Enrollment: 409 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2022-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (26):
- Portugal (5):
  - Centro Hospitalar de Entre Douro e Vouga, Santa Maria da Feira, Aveiro District
  - Hospital Beatriz Angelo, Loures, Lisbon District
  - Hospital do Espirito Santo de Evora, Evora
  - Centro Hospitalar Universitario Lisboa Norte - Hospital de Santa Maria, Lisbon
  - Hospital Distrital de Santarem, Santarém
- Spain (21):
  - Hospital Universitari Son Espases, Palma, Balearic Islands
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Canary Islands
  - Hospital Universitario de Leon, León, Castille and León
  - Hospital Universitario de Salamanca, Salamanca, Castille and León
  - Hospital Vall d'Hebron, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Universitari Parc Tauli, Barcelona, Catalonia
  - Hospital de Sant Joan Despi - Moises Broggi, Barcelona, Catalonia
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona, Catalonia
  - Hospital de La Princesa, Madrid, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid, Madrid
  - Hospital Clinico San Carlos, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario de La Paz, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid, Madrid
  - Hospital de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias (HUCA), Oviedo, Principality of Asturias
  - Hospital General Universitario de Alicante, Alicante, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario y Politecnico La Fe, Valencia, Valencia
  - Hospital de Manises, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Yarur A, Mantzaris GJ, Wang S, Adsul S, Kamble P, Cook E, Sajeev G, Guerin A, Bressler B. Stratified Patient Profiling for Vedolizumab Effectiveness in Crohn's Disease: Identifying Optimal Subgroups for Enhanced Treatment Response in the EVOLVE Study. Adv Ther. 2024 Jun;41(6):2324-2341. doi: 10.1007/s12325-024-02825-w. Epub 2024 Apr 24. PMID 38658485

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 25 investigative sites in Spain and Portugal from 19 February 2019 to 21 February 2022.
Pre-assignment Details: Participants diagnosed with Crohn's disease (CD) or ulcerative colitis (UC) and who initiated first or second line biologic treatment with vedolizumab or another biologic between January 2017 until date of site initiation were enrolled and observed retrospectively in this medical chart review study.
Groups:
- Cohort 1: Vedolizumab: Participants diagnosed with UC or CD, who had initiated first or second-line treatment with vedolizumab between January 2017 until date of site initiation (eligibility period) were observed in the pre-index event period from the date of UC or CD diagnosis until one day prior to the date of index vedolizumab treatment initiation during the eligibility period, and then in post-index event period from date of index vedolizumab treatment initiation until the earliest of 6 months (post-index treatment discontinuation, death of participant, lost-to-follow up, or date of chart abstraction). Index date was defined as the date when vedolizumab treatment was initiated.
- Cohort 2: Anti-TNF Alpha: Participants diagnosed with UC or CD, who had initiated first or second-line treatment with another biologic treatment (anti-tumour necrosis factor-alpha [TNF alpha]: infliximab, adalimumab, or golimumab [UC only]) between January 2017 until date of site initiation (eligibility period) were observed in the pre-index event period from the date of UC or CD diagnosis until one day prior to the date of index other biologic treatment initiation during the eligibility period, and then in post-index event period from date of index other biologic treatment initiation until the earliest of 6 months (post-index treatment discontinuation, death of participant, lost-to-follow up, or date of chart abstraction). Index date was defined as the date when other biologic treatment was initiated.
Period: Overall Study
Arm/Group | Cohort 1: Vedolizumab | Cohort 2: Anti-TNF Alpha
Started | 185 | 224
Completed | 172 | 212
Not Completed | 13 | 12
Not completed — Lost to Follow-up (at least 12 months) | 13 | 10
Not completed — Missing | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants with UC or CD that met all the inclusion criteria and none of exclusion were enrolled in this study.
Groups:
- Cohort 2: Anti-TNF Alpha: Participants diagnosed with UC or CD, who had initiated first or second-line treatment with another biologic treatment (TNF alpha: infliximab, adalimumab, or golimumab [UC only]) between January 2017 until date of site initiation (eligibility period) were observed in the pre-index event period from the date of UC or CD diagnosis until one day prior to the date of index other biologic treatment initiation during the eligibility period, and then in post-index event period from date of index other biologic treatment initiation until the earliest of 6 months (post-index treatment discontinuation, death of participant, lost-to-follow up, or date of chart abstraction). Index date was defined as the date when other biologic treatment was initiated.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Vedolizumab | Cohort 2: Anti-TNF Alpha | Total
Number analyzed (Participants) | 185 | 224 | 409
Age, Customized [Count of Participants; unit: Participants]
  18 to 92 Years | 185 | 224 | 409
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 85 | 166
  Male | 104 | 139 | 243
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 159 | 199 | 358
  Portugal | 26 | 25 | 51
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (Kg/m^2)] — Population: Here, "number analyzed" signifies participants for whom BMI data was available at the baseline.
  kilogram per square meter (Kg/m^2)
    number analyzed (Participants) | 143 | 176 | 319
    (all) | 24.8 (4.3) | 24.5 (4.0) | 24.6 (4.2)
Smoking Status [Count of Participants; unit: Participants] — Population: Here, "number analyzed" signifies participants for whom smoking status data was available at the baseline.
  Participants
    Never Smoked: number analyzed (Participants) | 161 | 214 | 375
    Never Smoked | 74 | 113 | 187
    Former Smoker: number analyzed (Participants) | 161 | 214 | 375
    Former Smoker | 61 | 66 | 127
    Current Smoker: number analyzed (Participants) | 161 | 214 | 375
    Current Smoker | 26 | 35 | 61
Treatment History for CD Participants [Count of Participants; unit: Participants] — Population: Here, "number analyzed" signifies CD participants for whom data for treatment history was available at the baseline.
  Participants
    Corticosteroids: number analyzed (Participants) | 69 | 115 | 184
    Corticosteroids | 37 | 61 | 98
    Immunomodulators: number analyzed (Participants) | 69 | 115 | 184
    Immunomodulators | 36 | 63 | 99
    Antibiotics: number analyzed (Participants) | 69 | 115 | 184
    Antibiotics | 7 | 17 | 24
    5-aminosalicylic acid (5-ASA): number analyzed (Participants) | 69 | 115 | 184
    5-aminosalicylic acid (5-ASA) | 28 | 34 | 62
    Other: number analyzed (Participants) | 69 | 115 | 184
    Other | 14 | 46 | 60
Treatment History for UC Participants [Count of Participants; unit: Participants] — Population: Here, "number analyzed" signifies UC participants for whom data for treatment history was available at the baseline.
  Participants
    Corticosteroids: number analyzed (Participants) | 96 | 94 | 190
    Corticosteroids | 57 | 66 | 123
    Corticosteroids Immunomodulators: number analyzed (Participants) | 96 | 94 | 190
    Corticosteroids Immunomodulators | 42 | 44 | 86
    Immunomodulators: number analyzed (Participants) | 96 | 94 | 190
    Immunomodulators | 4 | 8 | 12
    5-ASA: number analyzed (Participants) | 96 | 94 | 190
    5-ASA | 68 | 73 | 141
    Other: number analyzed (Participants) | 96 | 94 | 190
    Other | 25 | 27 | 52
Type of Inflammatory Bowel Disease (IBD) [Count of Participants; unit: Participants]
  CD | 83 | 127 | 210
  UC | 102 | 97 | 199
Age at First Ever CD Diagnosis [Mean (Standard Deviation); unit: years] — Population: Here, "number analyzed" signifies CD participants for whom data for age at first ever diagnosis was available at the baseline.
  years
    number analyzed (Participants) | 60 | 107 | 167
    (all) | 47.6 (17.3) | 35.0 (16.0) | 39.5 (17.5)
Age at First Ever UC diagnosis [Mean (Standard Deviation); unit: years] — Population: Here, "number analyzed" signifies UC participants for whom data for age at first ever diagnosis was available at the baseline.
  years
    number analyzed (Participants) | 78 | 76 | 154
    (all) | 44.6 (19.2) | 37.6 (14.8) | 41.1 (17.5)
Location of Intestinal Involvement at Diagnosis in CD Participants [Count of Participants; unit: Participants] — Population: Here, "number analyzed" signifies CD participants for whom data for location of intestinal involvement at diagnosis was available at the baseline.
  Participants
    Ileal: number analyzed (Participants) | 83 | 127 | 210
    Ileal | 51 | 53 | 104
    Colonic: number analyzed (Participants) | 83 | 127 | 210
    Colonic | 10 | 17 | 27
    Upper Gastrointestinal Tract: number analyzed (Participants) | 83 | 127 | 210
    Upper Gastrointestinal Tract | 8 | 13 | 21
    Ileocolonic: number analyzed (Participants) | 83 | 127 | 210
    Ileocolonic | 22 | 55 | 77
Location of UC at Diagnosis [Count of Participants; unit: Participants] — Population: Here, "number analyzed" signifies UC participants for whom data for location of UC diagnosis was available at the baseline.
  Participants
    Proctitis/proctosigmoiditis: number analyzed (Participants) | 98 | 92 | 190
    Proctitis/proctosigmoiditis | 23 | 17 | 40
    Left-sided (Distal to Splenic flexure): number analyzed (Participants) | 98 | 92 | 190
    Left-sided (Distal to Splenic flexure) | 35 | 31 | 66
    Extensive Colitis (Proximal to Hepatic Flexure): number analyzed (Participants) | 98 | 92 | 190
    Extensive Colitis (Proximal to Hepatic Flexure) | 40 | 44 | 84
Type of Active Fistulas at Diagnosis in CD Participants [Count of Participants; unit: Participants] — Population: Here, "number analyzed" signifies CD participants for whom data for type of active fistulas at diagnosis was available at the baseline.
  Participants
    Anal: number analyzed (Participants) | 7 | 24 | 31
    Anal | 3 | 17 | 20
    Rectovaginal: number analyzed (Participants) | 7 | 24 | 31
    Rectovaginal | 0 | 2 | 2
    Enterocutaneous: number analyzed (Participants) | 7 | 24 | 31
    Enterocutaneous | 2 | 2 | 4
    Internal: number analyzed (Participants) | 7 | 24 | 31
    Internal | 2 | 4 | 6
Type of Disease Behavior at Diagnosis Inflammatory in CD Participants [Count of Participants; unit: Participants] — Population: Here, "number analyzed" signifies CD participants for whom data for type of disease behavior at diagnosis inflammatory was available at the baseline.
  Participants
    Inflammatory: number analyzed (Participants) | 79 | 120 | 199
    Inflammatory | 37 | 74 | 111
    Stricturing: number analyzed (Participants) | 79 | 120 | 199
    Stricturing | 36 | 35 | 71
    Penetrating: number analyzed (Participants) | 79 | 120 | 199
    Penetrating | 9 | 19 | 28
    Anal: number analyzed (Participants) | 79 | 120 | 199
    Anal | 2 | 12 | 14
Participants With and Without Active Fistulas at Diagnosis in CD Participants [Count of Participants; unit: Participants] — Population: Here, "number analyzed" signifies CD participants for whom data for active fistulas at diagnosis was available at the baseline.
  Participants
    Participants with Active Fistulas at Diagnosis in CD Participants: number analyzed (Participants) | 75 | 107 | 182
    Participants with Active Fistulas at Diagnosis in CD Participants | 8 | 27 | 35
    Participants Without Active Fistulas at Diagnosis in CD Participants: number analyzed (Participants) | 75 | 107 | 182
    Participants Without Active Fistulas at Diagnosis in CD Participants | 67 | 80 | 147
Number of Fistulas in CD Participants [Mean (Standard Deviation); unit: number of fistulas] — Population: Here, "number analyzed" signifies CD participants for whom data for number of fistulas at diagnosis was available at the baseline.
  number of fistulas
    number analyzed (Participants) | 7 | 19 | 26
    (all) | 1.4 (0.8) | 1.2 (0.4) | 1.3 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With One or More Treatment Intensifications for CD Participants
Description: Index treatment is the first or second line treatment with vedolizumab or other biologics. Index date was defined as the date when vedolizumab or other biologic treatment was initiated. Dose intensification was performed by shortening the interval between doses in most cases in all the subgroups.
Time Frame: From the date of diagnosis of CD (within previous 2 years) including index date until post-index treatment discontinuation, death, loss to follow up, or date of chart abstraction initiation (approximately 6 months post index date)
Population: All participants with CD that met all the inclusion criteria and none of exclusion were enrolled in this study.
Measure: Number; unit: percentage of participants
Groups:
- Cohort 1, CD Participants: Vedolizumab: Participants diagnosed with CD, who had initiated first or second-line treatment with vedolizumab between January 2017 until date of site initiation (eligibility period) were observed in the pre-index event period from the date of CD diagnosis until one day prior to the date of index vedolizumab treatment initiation during the eligibility period, and then in post-index event period from date of index vedolizumab treatment initiation until the earliest of 6 months (post-index treatment discontinuation, death of participant, lost-to-follow up, or date of chart abstraction). Index date was defined as the date when vedolizumab treatment was initiated.
- Cohort 2, CD Participants: Anti-TNF Alpha: Participants diagnosed with CD, who had initiated first or second-line treatment with another biologic treatment (TNF alpha: infliximab, adalimumab), between January 2017 until date of site initiation (eligibility period) were observed in the pre-index event period from the date of CD diagnosis until one day prior to the date of index other biologic treatment initiation during the eligibility period, and then in post-index event period from date of index other biologic treatment initiation until the earliest of 6 months (post-index treatment discontinuation, death of participant, lost-to-follow up, or date of chart abstraction). Index date was defined as the date when other biologic treatment was initiated.
Arm/Group | Cohort 1, CD Participants: Vedolizumab | Cohort 2, CD Participants: Anti-TNF Alpha
Number analyzed (Participants) | 83 | 127
percentage of participants | 30.7 | 42.1
Statistical Analysis 1: Comparison: Cohort 1, CD Participants: Vedolizumab vs Cohort 2, CD Participants: Anti-TNF Alpha; Test type: Superiority; p = 0.13202, Regression, Logistic; p-value was estimated with a logistic regression adjusted by propensity scores inverse probability treatment weighting (PS-IPTW); Odds Ratio (OR) = 0.61, 95% CI 2-sided [0.32 to 1.16] — Estimated with a logistic regression adjusted by PS-IPTW

2. Primary Outcome: Percentage of Participants With One or More Treatment Intensifications for UC Participants
Description: as for outcome 1
Time Frame: From the date of diagnosis of UC (within previous 2 years) including index date until post-index treatment discontinuation, death, loss to follow up, or date of chart abstraction initiation (approximately 6 months post index date)
Population: All participants with UC that met all the inclusion criteria and none of exclusion were enrolled in this study.
Measure: Number; unit: percentage of participants
Groups:
- Cohort 1, UC Participants: Vedolizumab: Participants diagnosed with UC, who had initiated first or second-line treatment with vedolizumab between January 2017 until date of site initiation (eligibility period) were observed in the pre-index event period from the date of UC diagnosis until one day prior to the date of index vedolizumab treatment initiation during the eligibility period, and then in post-index event period from date of index vedolizumab treatment initiation until the earliest of 6 months (post-index treatment discontinuation, death of participant, lost-to-follow up, or date of chart abstraction). Index date was defined as the date when vedolizumab treatment was initiated.
- Cohort 2, UC Participants: Anti-TNF Alpha: Participants diagnosed with UC, who had initiated first or second-line treatment with other biologic treatment (anti-TNF alpha: infliximab, adalimumab, or golimumab) between January 2017 until date of site initiation (eligibility period) were observed in the pre-index event period from the date of UC diagnosis until one day prior to the date of index other biologic treatment initiation during the eligibility period, and then in post-index event period from date of index other biologic treatment initiation until the earliest of 6 months (post-index treatment discontinuation, death of participant, lost-to-follow up, or date of chart abstraction). Index date was defined as the date when other biologic treatment was initiated.
Arm/Group | Cohort 1, UC Participants: Vedolizumab | Cohort 2, UC Participants: Anti-TNF Alpha
Number analyzed (Participants) | 102 | 97
percentage of participants | 43.5 | 39.5
Statistical Analysis 1: Comparison: Cohort 1, UC Participants: Vedolizumab vs Cohort 2, UC Participants: Anti-TNF Alpha; Test type: Superiority; p = 0.5861, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.65 to 2.13] — Estimated with a logistic regression adjusted by PS-IPTW

3. Primary Outcome: Number of Participants With Reasons for Treatment Modifications in CD Participants
Description: Index date was defined as the date when vedolizumab or other biologic treatment was initiated.
Time Frame: as for outcome 1
Population: All participants with CD that met all the inclusion criteria and none of exclusion were enrolled in this study. Here, "overall number of participants analyzed" signified those participants who were evaluable for this outcome measure and "number analyzed" signified participants who were evaluable for specified categories of this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, CD Participants: Vedolizumab | Cohort 2, CD Participants: Anti-TNF Alpha
Number analyzed (Participants) | 17 | 38
Participants
  Participants discontinued treatment in first-line group: Absence of primary response | 6 | 6
  Participants discontinued treatment in first-line group: Lost of response | 2 | 13
  Participants discontinued treatment in first-line group: Partial response | 2 | 3
  Participants discontinued treatment in first-line group: Adverse event | 4 | 10
  Participants discontinued treatment in first-line group: Remission | 0 | 1
  Participants discontinued treatment in first-line group: Other reasons | 3 | 5
  Participants discontinued treatment in first-line group: Missing | 0 | 0
  Participants discontinued treatment in second-line group: number analyzed (Participants) | 9 | 20
  Participants discontinued treatment in second-line group: Absence of primary response | 6 | 2
  Participants discontinued treatment in second-line group: Lost of response | 1 | 7
  Participants discontinued treatment in second-line group: Partial response | 0 | 1
  Participants discontinued treatment in second-line group: Adverse event | 0 | 6
  Participants discontinued treatment in second-line group: Remission | 0 | 0
  Participants discontinued treatment in second-line group: Other reasons | 2 | 4
  Participants discontinued treatment in second-line group: Missing | 0 | 0

4. Primary Outcome: Number of Participants With Reasons for Treatment Modifications in UC Participants
Description: Index date was defined as the date when vedolizumab or other biologic treatment was initiated.
Time Frame: as for outcome 2
Population: All participants with UC that met all the inclusion criteria and none of exclusion were enrolled in this study. Here, "overall number of participants analyzed" signified those participants who were evaluable for this outcome measure and "number analyzed" signified participants who were evaluable for specified categories of this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1, UC Participants: Vedolizumab | Cohort 2, UC Participants: Anti-TNF Alpha
Number analyzed (Participants) | 19 | 29
Participants
  Participants discontinued treatment in first-line group: Absence of primary response | 8 | 9
  Participants discontinued treatment in first-line group: Lost of response | 6 | 6
  Participants discontinued treatment in first-line group: Partial response | 0 | 2
  Participants discontinued treatment in first-line group: Adverse event | 0 | 3
  Participants discontinued treatment in first-line group: Remission | 0 | 3
  Participants discontinued treatment in first-line group: Other reasons | 4 | 6
  Participants discontinued treatment in first-line group: Missing | 1 | 0
  Participants discontinued treatment in second-line group: number analyzed (Participants) | 13 | 15
  Participants discontinued treatment in second-line group: Absence of primary response | 3 | 2
  Participants discontinued treatment in second-line group: Lost of response | 5 | 8
  Participants discontinued treatment in second-line group: Partial response | 1 | 3
  Participants discontinued treatment in second-line group: Adverse event | 1 | 0
  Participants discontinued treatment in second-line group: Remission | 1 | 1
  Participants discontinued treatment in second-line group: Other reasons | 2 | 1
  Participants discontinued treatment in second-line group: Missing | 0 | 0

5. Primary Outcome: Percentage of Participants Who Discontinued Index Therapy for CD Participants
Description: Index treatment is defined as the first or second line treatment with vedolizumab or other biologics. Index date was defined as the date when vedolizumab or other biologic treatment was initiated.
Time Frame: as for outcome 1
Population: All participants with CD that met all the inclusion criteria and none of exclusion were enrolled in this study.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, CD Participants: Vedolizumab | Cohort 2, CD Participants: Anti-TNF Alpha
Number analyzed (Participants) | 83 | 127
percentage of participants | 38.8 | 49.3
Statistical Analysis 1: Comparison: Cohort 1, CD Participants: Vedolizumab vs Cohort 2, CD Participants: Anti-TNF Alpha; Test type: Superiority; p = 0.1648, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.35 to 1.19] — Estimated with a logistic regression adjusted by PS-IPTW

6. Primary Outcome: Percentage of Participants Who Discontinued Index Therapy for UC Participants
Description: as for outcome 5
Time Frame: as for outcome 2
Population: All participants with UC that met all the inclusion criteria and none of exclusion were enrolled in this study.
Measure: Number; unit: percentage of participants
Groups:
- Cohort 2, UC Participants: Anti-TNF Alpha: Participants diagnosed with UC, who had initiated first or second-line treatment with another biologic treatment (TNF alpha: infliximab, adalimumab, golimumab), between January 2017 until date of site initiation (eligibility period) were observed in the pre-index event period from the date of UC diagnosis until one day prior to the date of index other biologic treatment initiation during the eligibility period, and then in post-index event period from date of index other biologic treatment initiation until the earliest of 6 months (post-index treatment discontinuation, death of participant, lost-to-follow up, or date of chart abstraction). Index date was defined as the date when other biologic treatment was initiated.
Arm/Group | Cohort 1, UC Participants: Vedolizumab | Cohort 2, UC Participants: Anti-TNF Alpha
Number analyzed (Participants) | 102 | 97
percentage of participants | 39.6 | 50.0
Statistical Analysis 1: Comparison: Cohort 1, UC Participants: Vedolizumab vs Cohort 2, UC Participants: Anti-TNF Alpha; Test type: Superiority; p = 0.1732, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.36 to 1.20] — Estimated with a logistic regression adjusted by PS-IPTW

7. Primary Outcome: Number of Participants Who Discontinue Index Treatment in Vedolizumab Cohort and Initiated Second-line Biologic Within 6 Months Post-index Treatment Discontinuation
Description: as for outcome 5
Time Frame: From the date of diagnosis of CD or UC (within previous 2 years) including index date until post-index treatment discontinuation, death, loss to follow up, or date of chart abstraction initiation (approximately 6 months post index date)
Population: All participants with UC or CD that met all the inclusion criteria and none of exclusion were enrolled in this study. Here, "overall number of participants analyzed" signified those participants who were evaluable for this outcome measure. This outcome measure was planned to be assessed only for Cohort 1: Vedolizumab group.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: CD Participants, Vedolizumab: Participants diagnosed with CD, who had initiated first or second-line treatment with vedolizumab between January 2017 until date of site initiation (eligibility period) were observed in the pre-index event period from the date of CD diagnosis until one day prior to the date of index vedolizumab treatment initiation during the eligibility period, and then in post-index event period from date of index vedolizumab treatment initiation until the earliest of 6 months (post-index treatment discontinuation, death of participant, lost-to-follow up, or date of chart abstraction). Index date was defined as the date when vedolizumab treatment was initiated.
- Cohort 1: UC Participants, Vedolizumab: Participants diagnosed with UC, who had initiated first or second-line treatment with vedolizumab between January 2017 until date of site initiation (eligibility period) were observed in the pre-index event period from the date of UC diagnosis until one day prior to the date of index vedolizumab treatment initiation during the eligibility period, and then in post-index event period from date of index vedolizumab treatment initiation until the earliest of 6 months (post-index treatment discontinuation, death of participant, lost-to-follow up, or date of chart abstraction). Index date was defined as the date when vedolizumab treatment was initiated.
Arm/Group | Cohort 1: CD Participants, Vedolizumab | Cohort 1: UC Participants, Vedolizumab
Number analyzed (Participants) | 26 | 31
Participants | 20 | 16

8. Primary Outcome: Time to Switching for Vedolizumab Participants
Description: Time to switching was defined as time from index treatment initiation until a participant initiated another biologic treatment (Vedolizumab, infliximab, adalimumab, or golimumab [UC only], tofacitinib, certolizumab and ustekinumab). Index treatment is defined as the first or second line treatment with vedolizumab or other biologics. Index date was defined as the date when vedolizumab or other biologic treatment was initiated.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Cohort 1: CD Participants, Vedolizumab | Cohort 1: UC Participants, Vedolizumab
Number analyzed (Participants) | 20 | 16
months | 11.29 [6.49 to 14.23] | 8.62 [6.55 to 16.16]

9. Primary Outcome: Time to Discontinuation for CD Participants
Description: Time to discontinuation was defined as time from index treatment initiation until participant discontinued index treatment without switching to another biologic therapy. Time to discontinuation was estimated with Kaplan-Meier method adjusted by PS-IPTW. Index treatment is defined as the first or second line treatment with vedolizumab or other biologics. Index date was defined as the date when vedolizumab or other biologic treatment was initiated.
Time Frame: as for outcome 1
Population: All participants with CD that met all the inclusion criteria and none of exclusion were enrolled in this study. Here, "overall number of participants analyzed" signified those participants who were evaluable for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Cohort 1, CD Participants: Vedolizumab | Cohort 2, CD Participants: Anti-TNF Alpha
Number analyzed (Participants) | 26 | 58
months | 7.1 [5.6 to 12.5] | 10.7 [7.1 to 20.2]
Statistical Analysis 1: Comparison: Cohort 1, CD Participants: Vedolizumab vs Cohort 2, CD Participants: Anti-TNF Alpha; CD: Vedolizumab Versus Other Biological; Test type: Superiority; p = 0.2011, Log Rank Test Adjusted by PS-IPTW; p-value was estimated with Log Rank test adjusted by PS-IPTW. Multiple Imputation has been performed to estimate PS-IPTW

10. Primary Outcome: Time to Discontinuation for UC Participants
Description: as for outcome 9
Time Frame: as for outcome 2
Population: All participants with UC that met all the inclusion criteria and none of exclusion were enrolled in this study. Here, "overall number of participants analyzed" signified those participants who were evaluable for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Cohort 1, UC Participants: Vedolizumab | Cohort 2, UC Participants: Anti-TNF Alpha
Number analyzed (Participants) | 32 | 44
months | 9.0 [6.1 to 15.6] | 10.1 [5.7 to 15.2]
Statistical Analysis 1: Comparison: Cohort 1, UC Participants: Vedolizumab vs Cohort 2, UC Participants: Anti-TNF Alpha; Test type: Superiority; p = 0.6939, Log Rank Test Adjusted by PS-IPTW; [statistical method as in outcome 9, analysis 1]

11. Primary Outcome: Percentage of Participants With Clinical Response at 14 Weeks for CD Participants
Description: Clinical response in CD participants was evaluated using Harvey-Bradshaw index (HBI) scale. HBI scale consisted of clinical parameters: general well-being (0-4, where higher score means lower wellbeing), abdominal pain (0-3, higher score means more severe pain), number of liquid stools per day, abdominal mass (0-3, where higher score means presence of swelling in the abdomen), and complications (score 1 per item). Total score was the sum of individual parameters. The score ranged from a minimum score of 0 to no pre-specified maximum score as it depended on the number of liquid stools, where higher scores indicated more severe disease. Clinical response was defined as HBI score less than or equal to (<=) 4 or reduction of greater than or equal to (>=) 3 points in scores from index date or based on physician assessment. Index date was defined as the date when vedolizumab or other biologic treatment was initiated.
Time Frame: At 14 weeks post-index (assessment time window 10 to 18 weeks)
Population: All participants with CD that met all the inclusion criteria and none of exclusion were enrolled in this study. Here, "overall number of participants analyzed" signified those participants who were evaluable for this outcome measure. As pre-specified in the statistical analysis plan (SAP), the data inside 10 to 18 weeks time window was considered for 14 weeks assessment and were reported in this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, CD Participants: Vedolizumab | Cohort 2, CD Participants: Anti-TNF Alpha
Number analyzed (Participants) | 62 | 94
percentage of participants | 68.1 [lower limit 4.1] | 88.2 [lower limit 3.7]
Statistical Analysis 1: Comparison: Cohort 1, CD Participants: Vedolizumab vs Cohort 2, CD Participants: Anti-TNF Alpha; Test type: Superiority; p = 0.0071, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 0.29, 95% CI 2-sided [0.12 to 0.71] — Estimated with a logistic regression adjusted by PS-IPTW

12. Primary Outcome: Percentage of Participants With Clinical Response at 52 Weeks for CD Participants
Description: Clinical response in CD participants was evaluated using HBI scale. HBI scale consisted of clinical parameters: general well-being (0-4, where higher score means lower wellbeing), abdominal pain (0-3, higher score means more severe pain), number of liquid stools per day, abdominal mass (0-3, where higher score means presence of swelling in the abdomen), and complications (score 1 per item). Total score was the sum of individual parameters. The score ranged from a minimum score of 0 to no pre-specified maximum score as it depended on the number of liquid stools, where higher scores indicated more severe disease. Clinical response was defined as HBI score of <=4 or reduction of >=3 points in scores from index date or based on physician assessment. Index date was defined as the date when vedolizumab or other biologic treatment was initiated.
Time Frame: At 52 weeks post-index (assessment time window 46 to 58 weeks)
Population: All participants with CD that met all the inclusion criteria and none of exclusion were enrolled in this study. Here, "overall number of participants analyzed" signified those participants who were evaluable for this outcome measure. As pre-specified in the SAP, the data inside 46 to 58 weeks time window was considered for 52 weeks assessment and were reported in this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, CD Participants: Vedolizumab | Cohort 2, CD Participants: Anti-TNF Alpha
Number analyzed (Participants) | 75 | 119
percentage of participants | 74.8 [lower limit 2.3] | 69.8 [lower limit 2.5]
Statistical Analysis 1: Comparison: Cohort 1, CD Participants: Vedolizumab vs Cohort 2, CD Participants: Anti-TNF Alpha; Test type: Superiority; p = 0.4809, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.64 to 2.55] — Estimated with a logistic regression adjusted by PS-IPTW

13. Primary Outcome: Percentage of Participants With Clinical Response at 14 Weeks for UC Participants
Description: Clinical response in UC participants was evaluated using partial mayo score. Partial mayo score consisted of 3 sub-scores: stool pattern, most severe rectal bleeding of the day, and global assessment by physician, each graded from 0 to 3. These scores were summed to give a total score range of 0 to 9. Where, higher scores indicate more severe disease. Clinical response was defined as partial mayo score of less than (<) 4 or reduction of >= 2 points in scores from index date or based on physician assessment. Index date was defined as the date when vedolizumab or other biologic treatment was initiated. As pre-specified in the SAP, the data inside 10 to 18 weeks time window was considered for 14 weeks assessment and were reported in this outcome measure.
Time Frame: At 14 weeks post-index (assessment time window 10 to 18 weeks)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, UC Participants: Vedolizumab | Cohort 2, UC Participants: Anti-TNF Alpha
Number analyzed (Participants) | 81 | 78
percentage of participants | 81.2 [lower limit 2.3] | 80.5 [lower limit 2.5]
Statistical Analysis 1: Comparison: Cohort 1, UC Participants: Vedolizumab vs Cohort 2, UC Participants: Anti-TNF Alpha; Test type: Superiority; p = 0.9150, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.46 to 2.36] — Estimated with a logistic regression adjusted by PS-IPTW

14. Primary Outcome: Percentage of Participants With Clinical Response at 52 Weeks for UC Participants
Description: Clinical response in UC participants was evaluated using partial mayo score. Partial mayo score consisted of 3 sub-scores: stool pattern, most severe rectal bleeding of the day, and global assessment by physician, each graded from 0 to 3. These scores were summed to give a total score range of 0 to 9. Where, higher scores indicate more severe disease. The clinical response was defined as partial mayo score of <4 or reduction of >= 2 points in scores from index date or based on physician assessment. Index date was defined as the date when vedolizumab or other biologic treatment was initiated. As pre-specified in the SAP, the data inside 46 to 58 weeks time window was considered for 52 weeks assessment and were reported in this outcome measure.
Time Frame: At 52 weeks post-index (assessment time window 46 to 58 weeks)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, UC Participants: Vedolizumab | Cohort 2, UC Participants: Anti-TNF Alpha
Number analyzed (Participants) | 93 | 93
percentage of participants | 75.6 [lower limit 7.3] | 73.2 [lower limit 6.0]
Statistical Analysis 1: Comparison: Cohort 1, UC Participants: Vedolizumab vs Cohort 2, UC Participants: Anti-TNF Alpha; Test type: Superiority; p = 0.7254, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.56 to 2.28] — Estimated with a logistic regression adjusted by PS-IPTW

15. Primary Outcome: Percentage of Participants With Clinical Remission at 14 Weeks for CD Participants
Description: Clinical remission in CD participants was evaluated using HBI scale. HBI scale consisted of clinical parameters: general well-being (0-4, where higher score means lower wellbeing), abdominal pain (0-3, higher score means more severe pain), number of liquid stools per day, abdominal mass (0-3, where higher score means presence of swelling in the abdomen), and complications (score 1 per item). Total score was the sum of individual parameters. The score ranged from a minimum score of 0 to no pre-specified maximum score as it depended on the number of liquid stools, where higher scores indicated more severe disease. Clinical remission was defined as HBI score of <=4 or based on physician assessment. Index date was defined as the date when vedolizumab or other biologic treatment was initiated. As pre-specified in the SAP, the data inside 10 to 18 weeks time window was considered for 14 weeks assessment and were reported in this outcome measure.
Time Frame: At 14 weeks post-index (assessment time window 10 to 18 weeks)
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, CD Participants: Vedolizumab | Cohort 2, CD Participants: Anti-TNF Alpha
Number analyzed (Participants) | 62 | 94
percentage of participants | 56.2 [lower limit 7.3] | 79.3 [lower limit 6.0]
Statistical Analysis 1: Comparison: Cohort 1, CD Participants: Vedolizumab vs Cohort 2, CD Participants: Anti-TNF Alpha; Test type: Superiority; p = 0.0051, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 0.34, 95% CI 2-sided [0.16 to 0.72] — Estimated with a logistic regression adjusted by PS-IPTW

16. Primary Outcome: Percentage of Participants With Clinical Remission at 52 Weeks for CD Participants
Description: Clinical remission in CD participants was evaluated using HBI scale. HBI scale consisted of clinical parameters: general well-being (0-4, where higher score means lower wellbeing), abdominal pain (0-3, higher score means more severe pain), number of liquid stools per day, abdominal mass (0-3, where higher score means presence of swelling in the abdomen), and complications (score 1 per item). Total score was the sum of individual parameters. The score ranged from a minimum score of 0 to no pre-specified maximum score as it depended on the number of liquid stools, where higher scores indicated more severe disease. Clinical remission was defined as HBI score of <=4 or based on physician assessment. Index date was defined as the date when vedolizumab or other biologic treatment was initiated. As pre-specified in the SAP, the data inside 46 to 58 weeks time window was considered for 52 weeks assessment and were reported in this outcome measure.
Time Frame: At 52 weeks post-index (assessment time window 46 to 58 weeks)
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, CD Participants: Vedolizumab | Cohort 2, CD Participants: Anti-TNF Alpha
Number analyzed (Participants) | 75 | 119
percentage of participants | 51.3 | 66.5
Statistical Analysis 1: Comparison: Cohort 1, CD Participants: Vedolizumab vs Cohort 2, CD Participants: Anti-TNF Alpha; Test type: Superiority; p = 0.0653, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 0.53, 95% CI 2-sided [0.27 to 1.04] — Estimated with a logistic regression adjusted by PS-IPTW

17. Primary Outcome: Percentage of Participants With Clinical Remission at 14 Weeks for UC Participants
Description: Clinical remission in UC participants was evaluated using partial mayo score. Partial mayo score consisted of 3 sub-scores: stool pattern, most severe rectal bleeding of the day, and global assessment by physician, each graded from 0 to 3. These scores were summed to give a total score range of 0 to 9. Where, higher scores indicate more severe disease. Clinical remission was defined as partial mayo score of <2 or based on physician assessment. Index date was defined as the date when vedolizumab or other biologic treatment was initiated. As pre-specified in the SAP, the data inside 10 to 18 weeks time window was considered for 14 weeks assessment and were reported in this outcome measure.
Time Frame: At 14 weeks post-index (assessment time window 10 to 18 weeks)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, UC Participants: Vedolizumab | Cohort 2, UC Participants: Anti-TNF Alpha
Number analyzed (Participants) | 81 | 78
percentage of participants | 52.2 | 54.7
Statistical Analysis 1: Comparison: Cohort 1, UC Participants: Vedolizumab vs Cohort 2, UC Participants: Anti-TNF Alpha; Test type: Superiority; p = 0.7629, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.47 to 1.74] — Estimated with a logistic regression adjusted by PS-IPTW

18. Primary Outcome: Percentage of Participants With Clinical Remission at 52 Weeks for UC Participants
Description: Clinical remission in UC participants was evaluated using partial mayo score. Partial mayo score consisted of 3 sub-scores: stool pattern, most severe rectal bleeding of the day, and global assessment by physician, each graded from 0 to 3. These scores were summed to give a total score range of 0 to 9. Where, higher scores indicate more severe disease. Clinical remission was defined as partial mayo score of <2 or based on physician assessment. Index date was defined as the date when vedolizumab or other biologic treatment was initiated. As pre-specified in the SAP, the data inside 46 to 58 weeks time window was considered for 52 weeks assessment and were reported in this outcome measure.
Time Frame: At 52 weeks post-index (assessment time window 46 to 58 weeks)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, UC Participants: Vedolizumab | Cohort 2, UC Participants: Anti-TNF Alpha
Number analyzed (Participants) | 93 | 93
percentage of participants | 56.6 | 62.0
Statistical Analysis 1: Comparison: Cohort 1, UC Participants: Vedolizumab vs Cohort 2, UC Participants: Anti-TNF Alpha; Test type: Superiority; p = 0.4895, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.43 to 1.50] — Estimated with a logistic regression adjusted by PS-IPTW

19. Primary Outcome: Percentage of Participants With Biochemical Remission Based on C-reactive Protein (CRP) at 14 Weeks for CD Participants
Description: Biochemical remission based on CRP was defined as CRP level of <5 milligram per liter (mg/L). Index date was defined as the date when vedolizumab or other biologic treatment was initiated. As pre-specified in the SAP, the data inside greater than (>) 0 to 38 weeks time window was considered for 14 weeks assessment and were reported in this outcome measure.
Time Frame: At 14 weeks post-index (assessment time window >0 to 38 weeks)
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, CD Participants: Vedolizumab | Cohort 2, CD Participants: Anti-TNF Alpha
Number analyzed (Participants) | 80 | 116
percentage of participants | 69.1 [lower limit 24.50] | 74.6 [lower limit 38.01]
Statistical Analysis 1: Comparison: Cohort 1, CD Participants: Vedolizumab vs Cohort 2, CD Participants: Anti-TNF Alpha; Test type: Superiority; p = 0.4458, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.38 to 1.54] — Estimated with a logistic regression adjusted by PS-IPTW

20. Primary Outcome: Percentage of Participants With Biochemical Remission Based on CRP at 52 Weeks for CD Participants
Description: Biochemical remission based on CRP was defined as CRP level of <5 mg/L. Index date was defined as the date when vedolizumab or other biologic treatment was initiated. As pre-specified in the SAP, the data inside 28 to 76 weeks time window was considered for 52 weeks assessment and were reported in this outcome measure.
Time Frame: At 52 weeks post-index (assessment time window 28 to 76 weeks)
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, CD Participants: Vedolizumab | Cohort 2, CD Participants: Anti-TNF Alpha
Number analyzed (Participants) | 70 | 110
percentage of participants | 72.9 [lower limit 24.50] | 73.4 [lower limit 38.01]
Statistical Analysis 1: Comparison: Cohort 1, CD Participants: Vedolizumab vs Cohort 2, CD Participants: Anti-TNF Alpha; Test type: Superiority; p = 0.9471, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.47 to 2.04] — Estimated with a logistic regression adjusted by PS-IPTW

21. Primary Outcome: Percentage of Participants With Biochemical Remission Based on CRP at 14 Weeks for UC Participants
Description: Biochemical remission based on CRP was defined as CRP level <5 mg/L. Index date was defined as the date when vedolizumab or other biologic treatment was initiated. As pre-specified in the SAP, the data inside >0 to 38 weeks time window was considered for 14 weeks assessment and were reported in this outcome measure.
Time Frame: At 14 weeks post-index (assessment time window >0 to 38 weeks)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, UC Participants: Vedolizumab | Cohort 2, UC Participants: Anti-TNF Alpha
Number analyzed (Participants) | 97 | 87
percentage of participants | 58.5 | 77.2
Statistical Analysis 1: Comparison: Cohort 1, UC Participants: Vedolizumab vs Cohort 2, UC Participants: Anti-TNF Alpha; Test type: Superiority; p = 0.0104, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 0.42, 95% CI 2-sided [0.21 to 0.81] — Estimated with a logistic regression adjusted by PS-IPTW

22. Primary Outcome: Percentage of Participants With Biochemical Remission Based on CRP at 52 Weeks for UC Participants
Description: as for outcome 20
Time Frame: At 52 weeks post-index (assessment time window 28 to 76 weeks)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, UC Participants: Vedolizumab | Cohort 2, UC Participants: Anti-TNF Alpha
Number analyzed (Participants) | 89 | 76
percentage of participants | 60.4 | 85.2
Statistical Analysis 1: Comparison: Cohort 1, UC Participants: Vedolizumab vs Cohort 2, UC Participants: Anti-TNF Alpha; Test type: Superiority; p = 0.0011, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 0.26, 95% CI 2-sided [0.12 to 0.59] — Estimated with a logistic regression adjusted by PS-IPTW

23. Primary Outcome: Percentage of Participants With Biochemical Remission Based on Fecal Calprotectin (FCP) at 14 Weeks for CD Participants
Description: Biochemical remission based on FCP was defined as FCP level of <250 microgram per gram (mcg/g). Index date was defined as the date when vedolizumab or other biologic treatment was initiated. As pre-specified in the SAP, the data inside >0 to 38 weeks time window was considered for 14 weeks assessment and were reported in this outcome measure.
Time Frame: At 14 weeks post-index (assessment time window >0 to 38 weeks)
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, CD Participants: Vedolizumab | Cohort 2, CD Participants: Anti-TNF Alpha
Number analyzed (Participants) | 70 | 110
percentage of participants | 72.9 [lower limit 26.57] | 73.4 [lower limit 23.86]
Statistical Analysis 1: Comparison: Cohort 1, CD Participants: Vedolizumab vs Cohort 2, CD Participants: Anti-TNF Alpha; CD Participants; Test type: Superiority; p = 0.9471, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.47 to 2.04] — Estimated with a logistic regression adjusted by PS-IPTW

24. Primary Outcome: Percentage of Participants With Biochemical Remission Based on FCP at 52 Weeks for CD Participants
Description: Biochemical remission based on FCP was defined as FCP level of <250 mcg/g. Index date was defined as the date when vedolizumab or other biologic treatment was initiated. As pre-specified in the SAP, the data inside 28 to 76 weeks time window was considered for 52 weeks assessment and were reported in this outcome measure.
Time Frame: At 52 weeks post-index (assessment time window 28 to 76 weeks)
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, CD Participants: Vedolizumab | Cohort 2, CD Participants: Anti-TNF Alpha
Number analyzed (Participants) | 44 | 59
percentage of participants | 45.7 [lower limit 26.57] | 73.4 [lower limit 23.86]
Statistical Analysis 1: Comparison: Cohort 1, CD Participants: Vedolizumab vs Cohort 2, CD Participants: Anti-TNF Alpha; Test type: Superiority; p = 0.0104, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 0.30, 95% CI 2-sided [0.12 to 0.75] — Estimated with a logistic regression adjusted by PS-IPTW

25. Primary Outcome: Percentage of Participants With Biochemical Remission Based on FCP at 14 Weeks for UC Participants
Description: Biochemical remission based on FCP was defined as FCP level of <250 mcg/g. Index date was defined as the date when vedolizumab or other biologic treatment was initiated. As pre-specified in the SAP, the data inside >0 to 38 weeks time window was considered for 14 weeks assessment and were reported in this outcome measure.
Time Frame: At 14 weeks post-index (assessment time window >0 to 38 weeks)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, UC Participants: Vedolizumab | Cohort 2, UC Participants: Anti-TNF Alpha
Number analyzed (Participants) | 89 | 76
percentage of participants | 60.4 | 85.2
Statistical Analysis 1: Comparison: Cohort 1, UC Participants: Vedolizumab vs Cohort 2, UC Participants: Anti-TNF Alpha; Test type: Superiority; p = 0.0011, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 0.26, 95% CI 2-sided [0.12 to 0.59] — Estimated with a logistic regression adjusted by PS-IPTW

26. Primary Outcome: Percentage of Participants With Biochemical Remission Based on FCP at 52 Weeks for UC Participants
Description: as for outcome 24
Time Frame: At 52 weeks post-index (assessment time window 28 to 76 weeks)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, UC Participants: Vedolizumab | Cohort 2, UC Participants: Anti-TNF Alpha
Number analyzed (Participants) | 66 | 53
percentage of participants | 59.7 | 53.7
Statistical Analysis 1: Comparison: Cohort 1, UC Participants: Vedolizumab vs Cohort 2, UC Participants: Anti-TNF Alpha; Test type: Superiority; p = 0.5400, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.59 to 2.78] — Estimated with a logistic regression adjusted by PS-IPTW

27. Primary Outcome: Percentage of Participants With Endoscopic Response at 52 Weeks for CD Participants
Description: Endoscopic response for CD participants was evaluated using simple endoscopic index for Crohn's disease (SES-CD) score. SES-CD evaluated 4 endoscopic variables (ulcer size, percentage of the surface area that was ulcerated, percentage of the surface area affected, and stenosis in 5 segments evaluated during ileocolonoscopy (ileum, right colon, transverse colon, left colon, and rectum). The score for each endoscopic variable was the sum of values obtained for each segment. The SES-CD total was the sum of the 4 endoscopic variable scores from 0 to 56, where higher scores indicate more severe disease. Endoscopic response was defined as SES-CD score <=2 or based on physician assessment (for UC and CD both). SES-CD score at index date >0 relative difference was calculated (100*[Index date-52 weeks assessment]/Index date) and relative difference of >= 50% was considered response. Index date was defined as the date when vedolizumab or other biologic treatment was initiated.
Time Frame: At 52 weeks post-index (assessment time window 28 to 76 weeks)
Population: All participants with CD that met all the inclusion criteria and none of exclusion were enrolled in this study. Here, "overall number of participants analyzed" signified those participants who were evaluable for this outcome measure. As pre-specified in the SAP, the data inside 28 to 76 weeks time window was considered for 52 weeks assessment and were reported in this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, CD Participants: Vedolizumab | Cohort 2, CD Participants: Anti-TNF Alpha
Number analyzed (Participants) | 16 | 28
percentage of participants | 69.7 | 65.7
Statistical Analysis 1: Comparison: Cohort 1, CD Participants: Vedolizumab vs Cohort 2, CD Participants: Anti-TNF Alpha; Test type: Superiority; p = 0.8123, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.26 to 5.66] — Estimated with a logistic regression adjusted by PS-IPTW

28. Primary Outcome: Percentage of Participants With Endoscopic Response at 52 Weeks for UC Participants
Description: Endoscopic response in UC participants is based on investigator assessment. Index date was defined as the date when vedolizumab or other biologic treatment was initiated. As pre-specified in the SAP, the data inside 28 to 76 weeks time window was considered for 52 weeks assessment and were reported in this outcome measure.
Time Frame: At 52 weeks post-index (assessment time window 28 to 76 weeks)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Vedolizumab | Cohort 2: Anti-TNF Alpha
Number analyzed (Participants) | 23 | 22
percentage of participants | 44.8 | 78.2
Statistical Analysis 1: Comparison: Cohort 1: Vedolizumab vs Cohort 2: Anti-TNF Alpha; Test type: Superiority; p = 0.0282, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 0.22, 95% CI 2-sided [0.06 to 0.85] — Estimated with a logistic regression adjusted by PS-IPTW

29. Primary Outcome: Percentage of Participants With Endoscopic Remission at 52 Weeks for CD Participants
Description: Endoscopic remission for CD participants was evaluated using SES-CD score. The SES-CD evaluated 4 endoscopic variables (ulcer size, percentage of the surface area that was ulcerated, percentage of the surface area affected, and stenosis in 5 segments evaluated during ileocolonoscopy (ileum, right colon, transverse colon, left colon, and rectum). The score for each endoscopic variable was the sum of values obtained for each segment. The SES-CD total was the sum of the 4 endoscopic variable scores from 0 to 56, where higher scores indicate more severe disease. Endoscopic remission was defined as SES-CD score <=2 or based on physician assessment. Index date was defined as the date when vedolizumab or other biologic treatment was initiated. As pre-specified in the SAP, the data inside 28 to 76 weeks time window was considered for 52 weeks assessment and were reported in this outcome measure.
Time Frame: At 52 weeks post-index (assessment time window 28 to 76 weeks)
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, CD Participants: Vedolizumab | Cohort 2, CD Participants: Anti-TNF Alpha
Number analyzed (Participants) | 19 | 28
percentage of participants | 43.5 | 40.5
Statistical Analysis 1: Comparison: Cohort 1, CD Participants: Vedolizumab vs Cohort 2, CD Participants: Anti-TNF Alpha; Test type: Superiority; p = 0.8584, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.29 to 4.36] — Estimated with a logistic regression adjusted by PS-IPTW

30. Primary Outcome: Percentage of Participants With Endoscopic Remission at 52 Weeks for UC Participants
Description: Endoscopic remission in UC participants is based on investigator assessment. Index date was defined as the date when vedolizumab or other biologic treatment was initiated. As pre-specified in the SAP, the data inside 28 to 76 weeks time window was considered for 52 weeks assessment and were reported in this outcome measure.
Time Frame: At 52 weeks post-index (assessment time window 28 to 76 weeks)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, UC Participants: Vedolizumab | Cohort 2, UC Participants: Anti-TNF Alpha
Number analyzed (Participants) | 23 | 22
percentage of participants | 35.5 | 36.6
Statistical Analysis 1: Comparison: Cohort 1, UC Participants: Vedolizumab vs Cohort 2, UC Participants: Anti-TNF Alpha; Test type: Superiority; p = 0.9474, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.24 to 3.78] — Estimated with a logistic regression adjusted by PS-IPTW

31. Secondary Outcome: Percentage of Participants With Adverse Events and Serious Adverse Events
Description: Index event period was defined as the period of time within which participants with UC or CD initiated first or second line treatment with vedolizumab or other biologic. The PS-IPTW method was used for balancing the cohorts. Percentage of participants determined after applying this method are reported in 'Adverse events' and 'Serious adverse events' categories in this outcome measure.
Time Frame: Index event period up to 6 months post-index treatment discontinuation
Population: All participants with UC or CD that met all the inclusion criteria and none of exclusion were enrolled in this study.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, CD Participants: Vedolizumab | Cohort 2, CD Participants: Anti-TNF Alpha | Cohort 1, UC Participants: Vedolizumab | Cohort 2, UC Participants: Anti-TNF Alpha
Number analyzed (Participants) | 83 | 127 | 102 | 97
percentage of participants
  Adverse event | 50.7 | 58.4 | 33.4 | 55.0
  Serious adverse event | 26.5 | 23.2 | 16.9 | 23.9
Statistical Analysis 1: Comparison: Cohort 1, CD Participants: Vedolizumab vs Cohort 2, CD Participants: Anti-TNF Alpha; Adverse event; Test type: Superiority; p = 0.3103, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.40 to 1.34] — The incidence comparison was estimated by using a logistic regression adjusted by PS-IPTW. Multiple Imputation has been performed to estimate PS-IPTW
Statistical Analysis 2: Comparison: Cohort 1, UC Participants: Vedolizumab vs Cohort 2, UC Participants: Anti-TNF Alpha; Adverse event; Test type: Superiority; p = 0.0045, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 0.41, 95% CI 2-sided [0.22 to 0.76] — [estimate comment as in outcome 31, analysis 1]
Statistical Analysis 3: Comparison: Cohort 1, CD Participants: Vedolizumab vs Cohort 2, CD Participants: Anti-TNF Alpha; Serious adverse event; Test type: Superiority; p = 0.6287, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.59 to 2.42] — [estimate comment as in outcome 31, analysis 1]
Statistical Analysis 4: Comparison: Cohort 1, UC Participants: Vedolizumab vs Cohort 2, UC Participants: Anti-TNF Alpha; Serious adverse event; Test type: Superiority; p = 0.2495, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.31 to 1.36] — [estimate comment as in outcome 31, analysis 1]

32. Secondary Outcome: Incidence Rate of Adverse Events and Serious Adverse Events
Description: Incidence rate was based on per 100 participants-year. Index event period was defined as the period of time within which participants with UC or CD initiated first or second line treatment with vedolizumab or other biologic.
Time Frame: Index event period up to 6 months post-index treatment discontinuation
Population: All participants with UC or CD that met all the inclusion criteria and none of exclusion were enrolled in this study.
Measure: Number; unit: events per 100 participant-years
Arm/Group | Cohort 1, CD Participants: Vedolizumab | Cohort 2, CD Participants: Anti-TNF Alpha | Cohort 1, UC Participants: Vedolizumab | Cohort 2, UC Participants: Anti-TNF Alpha
Number analyzed (Participants) | 83 | 127 | 102 | 97
events per 100 participant-years
  Adverse event | 8.53 [lower limit 98.6] | 9.53 [lower limit 187.8] | 8.83 [lower limit 112.5] | 10.64 [lower limit 133.5]
  Serious adverse event | 4.62 | 2.31 | 4.17 | 3.21
Statistical Analysis 1: Comparison: Cohort 1, CD Participants: Vedolizumab vs Cohort 2, CD Participants: Anti-TNF Alpha; Adverse event; Test type: Superiority; p = 0.4784, Poisson Regression; p-value was estimated with a Poisson regression including the following time adjusted by PS-IPTW; Risk Ratio (RR) = 0.89, 95% CI 2-sided [0.66 to 1.22] — The incidence rate comparison was estimated by using a Poisson regression adjusted by PS-IPTW. Multiple Imputation has been performed to estimate PS-IPTW
Statistical Analysis 2: Comparison: Cohort 1, UC Participants: Vedolizumab vs Cohort 2, UC Participants: Anti-TNF Alpha; Adverse event; Test type: Superiority; p = 0.2616, Poisson Regression; p-value was estimated with a Poisson regression including the following time adjusted by PS-IPTW; Risk Ratio (RR) = 0.83, 95% CI 2-sided [0.60 to 1.15] — [estimate comment as in outcome 32, analysis 1]
Statistical Analysis 3: Comparison: Cohort 1, CD Participants: Vedolizumab vs Cohort 2, CD Participants: Anti-TNF Alpha; Serious adverse event; Test type: Superiority; p = 0.0077, Poisson Regression; p-value was estimated with a Poisson regression including the following time adjusted by PS-IPTW; Risk Ratio (RR) = 2.01, 95% CI 2-sided [1.20 to 3.34] — [estimate comment as in outcome 32, analysis 1]
Statistical Analysis 4: Comparison: Cohort 1, UC Participants: Vedolizumab vs Cohort 2, UC Participants: Anti-TNF Alpha; Serious adverse event; Test type: Superiority; p = 0.3046, Poisson Regression; p-value was estimated with a Poisson regression including the following time adjusted by PS-IPTW; Risk Ratio (RR) = 1.30, 95% CI 2-sided [0.79 to 2.14] — [estimate comment as in outcome 32, analysis 1]

33. Secondary Outcome: Percentage of Participants With Related Treatment Adverse Events and Related Treatment Serious Adverse Events
Description: Index event period was defined as the period of time within which participants with UC or CD initiated first or second line treatment with vedolizumab or other biologic. Percentage of participants with treatment related adverse events and related treatment serious adverse events were reported.
Time Frame: Index event period up to 6 months post-index treatment discontinuation
Population: All participants with UC or CD that met all the inclusion criteria and none of exclusion were enrolled in this study.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, CD Participants: Vedolizumab | Cohort 2, CD Participants: Anti-TNF Alpha | Cohort 1, UC Participants: Vedolizumab | Cohort 2, UC Participants: Anti-TNF Alpha
Number analyzed (Participants) | 83 | 127 | 102 | 97
percentage of participants
  Adverse events related to treatment | 11.6 | 19.6 | 2.1 | 8.5
  Serious adverse events related to treatment | 2.3 | 5.5 | 0.8 | 0.5
Statistical Analysis 1: Comparison: Cohort 1, CD Participants: Vedolizumab vs Cohort 2, CD Participants: Anti-TNF Alpha; Adverse events related to treatment; Test type: Superiority; p = 0.1681, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.22 to 1.30] — [estimate comment as in outcome 31, analysis 1]
Statistical Analysis 2: Comparison: Cohort 1, UC Participants: Vedolizumab vs Cohort 2, UC Participants: Anti-TNF Alpha; Adverse events related to treatment; Test type: Superiority; p = 0.0645, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 0.23, 95% CI 2-sided [0.05 to 1.09] — [estimate comment as in outcome 31, analysis 1]
Statistical Analysis 3: Comparison: Cohort 1, CD Participants: Vedolizumab vs Cohort 2, CD Participants: Anti-TNF Alpha; Serious adverse events related to treatment; Test type: Superiority; p = 0.3145, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 0.38, 95% CI 2-sided [0.06 to 2.51] — [estimate comment as in outcome 31, analysis 1]
Statistical Analysis 4: Comparison: Cohort 1, UC Participants: Vedolizumab vs Cohort 2, UC Participants: Anti-TNF Alpha; Serious adverse events related to treatment; Test type: Superiority; p = 0.8197, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 1.49, 95% CI 2-sided [0.05 to 47.11] — [estimate comment as in outcome 31, analysis 1]

34. Secondary Outcome: Incidence Rate of Related Treatment Adverse Events and Related Treatment Serious Adverse Events
Description: Incidence rate was based on per 100 participant-year. Index event period was defined as the period of time within which participants with UC or CD initiated first or second line treatment with vedolizumab or other biologic.
Time Frame: Index event period up to 6 months post-index treatment discontinuation
Population: All participants with UC or CD that met all the inclusion criteria and none of exclusion were enrolled in this study.
Measure: Number; unit: events per 100 participant-years
Arm/Group | Cohort 1, CD Participants: Vedolizumab | Cohort 2, CD Participants: Anti-TNF Alpha | Cohort 1, UC Participants: Vedolizumab | Cohort 2, UC Participants: Anti-TNF Alpha
Number analyzed (Participants) | 83 | 127 | 102 | 97
events per 100 participant-years
  Adverse events related to treatment | 1.15 | 2.70 | 0.23 | 1.10
  Serious adverse events related to treatment | 0.29 | 0.53 | 0.09 | 0.06
Statistical Analysis 1: Comparison: Cohort 1, CD Participants: Vedolizumab vs Cohort 2, CD Participants: Anti-TNF Alpha; Adverse events related to treatment; Test type: Superiority; p = 0.0239, Poisson Regression; p-value was estimated with a Poisson regression including the following time adjusted by PS-IPTW; Risk Ratio (RR) = 0.43, 95% CI 2-sided [0.20 to 0.89] — [estimate comment as in outcome 32, analysis 1]
Statistical Analysis 2: Comparison: Cohort 1, UC Participants: Vedolizumab vs Cohort 2, UC Participants: Anti-TNF Alpha; Adverse events related to treatment; Test type: Superiority; p = 0.0373, Poisson Regression; p-value was estimated with a Poisson regression including the following time adjusted by PS-IPTW; Risk Ratio (RR) = 0.21, 95% CI 2-sided [0.05 to 0.91] — [estimate comment as in outcome 32, analysis 1]
Statistical Analysis 3: Comparison: Cohort 1, CD Participants: Vedolizumab vs Cohort 2, CD Participants: Anti-TNF Alpha; Serious adverse events related to treatment; Test type: Superiority; p = 0.4260, Poisson Regression; p-value was estimated with a Poisson regression including the following time adjusted by PS-IPTW; Risk Ratio (RR) = 0.54, 95% CI 2-sided [0.12 to 2.49] — [estimate comment as in outcome 32, analysis 1]
Statistical Analysis 4: Comparison: Cohort 1, UC Participants: Vedolizumab vs Cohort 2, UC Participants: Anti-TNF Alpha; Serious adverse events related to treatment; Test type: Superiority; p = 0.8012, Poisson Regression; Risk Ratio (RR) = 1.56, 95% CI 2-sided [0.05 to 48.44] — [estimate comment as in outcome 32, analysis 1]

35. Secondary Outcome: Percentage of Participants With Infections, Serious Infections and Malignancies
Description: Index event period was defined as the period of time within which participants with UC or CD initiated first or second line treatment with vedolizumab or other biologic. Percentage of participants with infections, serious infections and malignancies were reported.
Time Frame: Index event period up to 6 months post-index treatment discontinuation
Population: All participants with UC or CD that met all the inclusion criteria and none of exclusion were enrolled in this study.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, CD Participants: Vedolizumab | Cohort 2, CD Participants: Anti-TNF Alpha | Cohort 1, UC Participants: Vedolizumab | Cohort 2, UC Participants: Anti-TNF Alpha
Number analyzed (Participants) | 83 | 127 | 102 | 97
percentage of participants | 4.1 | 19.8 | 6.4 | 17.8
Statistical Analysis 1: Comparison: Cohort 1, CD Participants: Vedolizumab vs Cohort 2, CD Participants: Anti-TNF Alpha; Test type: Superiority; p = 0.0044, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 0.17, 95% CI 2-sided [0.05 to 0.58] — [estimate comment as in outcome 31, analysis 1]
Statistical Analysis 2: Comparison: Cohort 1, UC Participants: Vedolizumab vs Cohort 2, UC Participants: Anti-TNF Alpha; Test type: Superiority; p = 0.0215, Regression, Logistic; p-value was estimated with a logistic regression adjusted by PS-IPTW; Odds Ratio (OR) = 0.32, 95% CI 2-sided [0.12 to 0.84] — [estimate comment as in outcome 31, analysis 1]

36. Secondary Outcome: Incidence Rate of Infections, Serious Infections and Malignancies
Description: as for outcome 34
Time Frame: Index event period up to 6 months post-index treatment discontinuation
Population: All participants with UC or CD that met all the inclusion criteria and none of exclusion were enrolled in this study.
Measure: Number; unit: events per 100 participant-years
Groups:
- Cohort 2, UC Participants: Anti-TNF Alpha: Participants diagnosed with UC, who had initiated first or second-line treatment with other biologic (infliximab, adalimumab, or golimumab) between January 2017 until date of site initiation (eligibility period) were observed from the date of UC diagnosis until one day prior to the date of index other biologic treatment initiation during the eligibility period, and then from date of index other biologic treatment initiation until the earliest of 6 months (post-index treatment discontinuation, death of participant, lost-to-follow up, or date of chart abstraction). Index date was defined as the date when other biologic treatment was initiated.
Arm/Group | Cohort 1, CD Participants: Vedolizumab | Cohort 2, CD Participants: Anti-TNF Alpha | Cohort 1, UC Participants: Vedolizumab | Cohort 2, UC Participants: Anti-TNF Alpha
Number analyzed (Participants) | 83 | 127 | 102 | 97
events per 100 participant-years | 0.48 | 1.75 | 0.75 | 2.42
Statistical Analysis 1: Comparison: Cohort 1, CD Participants: Vedolizumab vs Cohort 2, CD Participants: Anti-TNF Alpha; Test type: Superiority; p = 0.0152, Poisson Regression; p-value was estimated with a Poisson regression including the following time adjusted by PS-IPTW; Risk Ratio (RR) = 0.27, 95% CI 2-sided [0.10 to 0.78] — [estimate comment as in outcome 32, analysis 1]
Statistical Analysis 2: Comparison: Cohort 1, UC Participants: Vedolizumab vs Cohort 2, UC Participants: Anti-TNF Alpha; Test type: Superiority; p = 0.8012, Poisson Regression; p-value was estimated with a Poisson regression including the following time adjusted by PS-IPTW; Risk Ratio (RR) = 1.56, 95% CI 2-sided [0.05 to 48.44] — [estimate comment as in outcome 32, analysis 1]

ADVERSE EVENTS:
Time Frame: Index event period up to 6 months post-index treatment discontinuation
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. The number of participants affected with non-serious adverse events and serious adverse events are reported as collected (statistically unprocessed data).
Arm/Group | Cohort 1, CD Participants: Vedolizumab | Cohort 2, CD Participants: Anti-TNF Alpha | Cohort 1, UC Participants: Vedolizumab | Cohort 2, UC Participants: Anti-TNF Alpha
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/127 | 9/102 | 3/97
Serious Adverse Events (participants affected / at risk) | 23/83 | 26/127 | 16/102 | 21/97
Other Adverse Events (participants affected / at risk) | 20/83 | 49/127 | 18/102 | 31/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, CD Participants: Vedolizumab (N=83) | Cohort 2, CD Participants: Anti-TNF Alpha (N=127) | Cohort 1, UC Participants: Vedolizumab (N=102) | Cohort 2, UC Participants: Anti-TNF Alpha (N=97)
Crohn's disease (Gastrointestinal disorders) | 3 | 2 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 3 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Duodenal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Inflammatory bowel disease (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ileocaecal resection (Surgical and medical procedures) | 2 | 0 | 0 | 0
Abdominal wall operation (Surgical and medical procedures) | 1 | 0 | 0 | 0
Cholecystectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0
Hospitalisation (Surgical and medical procedures) | 1 | 1 | 2 | 0
Ileectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0
Ileocolostomy (Surgical and medical procedures) | 1 | 0 | 0 | 0
Knee operation (Surgical and medical procedures) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 1 | 0 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 3 | 1 | 1
Condition aggravated (General disorders) | 4 | 1 | 0 | 3
Axial spondyloarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Surgery (Surgical and medical procedures) | 0 | 1 | 0 | 0
Eventration repair (Surgical and medical procedures) | 0 | 1 | 0 | 0
Sarcoidosis (Immune system disorders) | 0 | 1 | 0 | 0
Antinuclear antibody positive (Investigations) | 0 | 1 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 1
Wound evisceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Fistulotomy (Surgical and medical procedures) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Large intestine infection (Infections and infestations) | 0 | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Cytomegalovirus colitis (Infections and infestations) | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0
Angioplasty (Surgical and medical procedures) | 0 | 0 | 1 | 0
Debridement (Surgical and medical procedures) | 0 | 0 | 1 | 0
Hernia repair (Surgical and medical procedures) | 0 | 0 | 1 | 0
Ileostomy (Surgical and medical procedures) | 0 | 0 | 1 | 0
Prostatectomy (Surgical and medical procedures) | 0 | 0 | 1 | 0
Sigmoidectomy (Surgical and medical procedures) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0
Biopsy colon (Investigations) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Superficial vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, CD Participants: Vedolizumab (N=83) | Cohort 2, CD Participants: Anti-TNF Alpha (N=127) | Cohort 1, UC Participants: Vedolizumab (N=102) | Cohort 2, UC Participants: Anti-TNF Alpha (N=97)
Crohn's disease (Gastrointestinal disorders) | 3 | 8 | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 3 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Furuncle (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 4 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0
Liver function test increased (Investigations) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 5 | 7
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 3 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 2 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 2
Pelvic abscess (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Salmonellosis (Infections and infestations) | 0 | 1 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Paradoxical psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 0 | 3 | 0 | 1
Asthenia (General disorders) | 0 | 4 | 1 | 3
Condition aggravated (General disorders) | 0 | 1 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0 | 0
Drug tolerance decreased (General disorders) | 0 | 1 | 0 | 0
Inflammation (General disorders) | 0 | 1 | 0 | 1
Oedema (General disorders) | 0 | 1 | 0 | 0
Polyp (General disorders) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Ejaculation disorder (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Dystonia (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0 | 0
Hyperferritinaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0
H1n1 influenza (Infections and infestations) | 0 | 0 | 1 | 0
Keratouveitis (Infections and infestations) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0
Secretion discharge (General disorders) | 0 | 0 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Delivery (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mass (General disorders) | 0 | 0 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1
Molluscum contagiosum (Infections and infestations) | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Eventration repair (Surgical and medical procedures) | 0 | 0 | 0 | 1
Lipids abnormal (Investigations) | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-05-23): https://cdn.clinicaltrials.gov/large-docs/86/NCT03710486/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-17): https://cdn.clinicaltrials.gov/large-docs/86/NCT03710486/SAP_001.pdf